CLINICAL TRIAL: NCT01375595
Title: The Role of the Inferior Frontal Gyrus in Long-Term Auditory Memory a rTMS Study
Brief Title: Brain Areas Involved in Sound and Spoken Word Memory
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110182; 11-N-0182
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2015-10-30

CONDITIONS: Brain Mapping; Language Disorder; Adult; Healthy; Memory Disorder
Keywords: Working Memory; Repetitive TMS (rTMS); Language; Healthy Volunteer; HV
MeSH Terms: conditions — Language Disorders; Memory Disorders; Language

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Studies have shown that animals such as monkeys and dogs have excellent sight and touch memory but perform poorly on sound memory tasks. Human brains have certain areas that are important for speaking and understanding language. These areas may be involved in sound and spoken word memory. Researchers want to study these areas of the brain to find out if the memory for sounds requires brain structures that are usually associated with language learning and are unique to humans.

Objectives:

- To use magnetic resonance imaging to study areas of the brain involved in sound memory.

Eligibility:

- Healthy right-handed volunteers between 18 and 50 years of age. They must be native English speakers and have completed high school.

Design:

* The study requires a screening visit and 1 or 2 study visits to the National Institutes of Health Clinical Center.
* At the screening visit, volunteers will have a medical history taken. They will also have physical and neurological exams, and complete a questionnaire. Women of childbearing age will give a urine sample. Participants who have not had a magnetic resonance imaging (MRI) scan in the past year will have one at this visit.
* At the second visit, participants will have tests of sound memory. They will listen to a set of nonsense words spoken through earphones and memorize the words. Then they will listen to the words again to judge if the words were part of the earlier list. Participants will have a 1 hour break, then do the sound memory test again. During the second test they will have repetitive transcranial magnetic stimulation (rTMS), which stimulates different regions of the brain.
* If the group results from the testing sessions are positive, there will be a third visit. At this visit, participants will have a sound perception test. They will listen to words spoken through earphones and judge whether the words in the pair are the same or different. Participants will have rTMS during these tests as well.

DETAILED DESCRIPTION:
Objective:

Humans are the only animals that use language to communicate with each other. Among many other requirements, humans need excellent auditory long-term memory to be able to master the complicated task of learning a language. It is still not completely understood which brain regions are involved in transferring auditory stimuli into long-term memory. The goal of this research proposal is to examine whether brain structures that are known to be essential in language production also play an important role in encoding auditory stimuli into long-term memory.

Study population:

We propose using repetitive transcranial magnetic stimulation (rTMS) to examine the role of

frontal and temporo-parietal cortical areas in the storage of auditory stimuli in long-term memory. The whole study will comprise three experiments. Each of the three experiments will consist of one to three sessions. Sessions 1 and 2 will be compulsory in every experiment. Session 3 will only be required if positive results are obtained in session 2. Every participant can only participate in one of the three planned experiments.

In Experiment 1, we will investigate the potential role of Broca s area in auditory memory. If we find that rTMS in Broca s area interferes with performance on the memory task, we will conduct a control (session 3) to determine whether or not the impairment was actually due to interference with stimulus perception rather than with memory, per se. We will conduct Experiment 2 to investigate the possible role of Wernicke s region in auditory memory. We will conduct Experiment 3 to investigate the role of the ventral premotor cortex (PMv) in auditory memory.

In experiment 2 and 3 we will also conduct the same control session 3, as in Experiment 1 if the rTMS impairs performance on the auditory memory task. All experiments will consist of two sessions and an additional, third session if rTMS-induced impairment is found. In that case all participants will be called back for the control experiment. During session 1, a neurological examination will be performed and a clinical, anatomical, and functional MRI (Magnetic Resonance Imaging) will be taken (functional MRI for second repeat of experiment 1 and for experiment 3). In session 2, rTMS will be used in an attempt to temporarily disrupt the function of Broca s area (experiment 1), the TPJ (experiment 2) or PMv (experiment 3) while participants are performing an auditory recognition memory task. By temporarily disrupting cortical functioning in those localized regions, we will be able to determine whether or not their function is crucial for encoding auditory stimuli into long-term memory. In the control session, to be conducted only if the experimental task yields a positive result (i.e., impairment), we will test auditory perception by asking participants to make same/different judgments on stimulus pairs (similar to those used in session 2) presented with a very short delay while using the same rTMS routine as in session 2.

By amendment, we wish to expand session 1 to include functional MRI (fMRI) imaging designed to identify and refine the targets for disruption by rTMS in the subsequent session: Broca s area (experiment 1), and PMv (experiment 3). Specifically, we intend to (1) repeat Experiment 1 of the approved protocol using fMRI localization in an additional 15 subjects, and (2) proceed with Experiment 3 as described in the original protocol, also with the addition of fMRI localization. Initial results in experiment 1 (Broca s area) fell just short of significance, possibly because anatomical landmarks are inconsistent between subjects (e.g., Amunts et al., 1999); an fMRI localizer in each subject could reduce this variability. Unlike in the previous protocol, session 1 can not be skipped if the subject has had a neurological exam and MRI in the past year (the exam may be skipped, but all subjects will need the fMRI). The maximum number of sessions per experiment will remain unchanged at three: 1) intake exam and anatomical/functional MRI, 2) rTMS, and 3) a control session only if a significant effect of rTMS is observed.

By amendment, we also wish to consider the three experiments to be independent, rather than each contingent on the outcome of the previous experiment(s). As outlined below (sections 2.3-2.5), experimental evidence implicates all three regions in the auditory-motor network under study. Preliminary evidence indicates a positive effect in experiment 2 (the TPJ), but this does not render experiment 3 moot. Therefore we wish to apply fMRI-targeted rTMS to Broca s area, and PMv, in independent experiments.

Outcome measures:

In session 2, the primary outcome measure will be the number of correctly remembered auditory stimuli. Secondary output will be reaction time during the recognition phase of the experiment.

In the control experiment (if conducted) the primary outcome measure will be the number of correct same/different judgments and, again, reaction time will be the secondary measure.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for this research study participants must:

Be between the ages of 18 and 50 years of age

Be free of any neurologic condition that might affect performance of the tasks in these experiments

Be right handed

Be native English speakers

Have a finished high-school education or equivalent, such as GED

EXCLUSION CRITERIA:

Participants will be excluded from this research study if they:

Are taking medications that include antidepressants, anxiolytics, anticonvulsants, antipsychotics, antiparkinson, hypnotics, stimulants, and/or antihistamines

Have a diagnosed neurologic or psychiatric condition

Have a history of seizure disorder

Have implanted devices such as pacemakers, medication pumps, or defibrillators, metal in the cranium except the mouth, intracardiac lines, history of shrapnel injury or any other condition/device that may contraindicate or preclude the acquisition of MRI

Have severe back pain or any other condition which might prevent them from lying flat for up to 1 hour

Have Claustrophobia (a fear of tight spaces), which prevents them from lying still in a tight or small space for up to 1 hour

Are currently pregnant

Have known hearing loss

Have an alcohol or substance abuse problem as determined by the screening we will do

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-05-26; Study Completion 2015-10-30

PRIMARY OUTCOMES:
The primary outcome of this study is the error rate during the recognition memory task. The error rate is defined by the amount of stimuli that are correctly classified as familiar or unfamiliar.

SECONDARY OUTCOMES:
The secondary outcome measure of this study is the reaction time of participants to make judgments concerning the familiarity during the recognition memory task.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aggleton JP, Brown MW. Interleaving brain systems for episodic and recognition memory. Trends Cogn Sci. 2006 Oct;10(10):455-63. doi: 10.1016/j.tics.2006.08.003. Epub 2006 Aug 28. PMID 16935547
- [Background] Andoh J, Artiges E, Pallier C, Riviere D, Mangin JF, Cachia A, Plaze M, Paillere-Martinot ML, Martinot JL. Modulation of language areas with functional MR image-guided magnetic stimulation. Neuroimage. 2006 Jan 15;29(2):619-27. doi: 10.1016/j.neuroimage.2005.07.029. Epub 2005 Sep 15. PMID 16168674
- [Background] Alloway TP, Alloway RG. Investigating the predictive roles of working memory and IQ in academic attainment. J Exp Child Psychol. 2010 May;106(1):20-9. doi: 10.1016/j.jecp.2009.11.003. Epub 2009 Dec 16. PMID 20018296